CLINICAL TRIAL: NCT01728480
Title: A Phase I Study of CBLB502 in the Treatment of Patients With Poor Prognosis Advanced Squamous Cell Carcinomas of the Head and Neck Receiving Chemoradiotherapy
Brief Title: Entolimod in Treating Patients With Stage III-IV Squamous Cell Head and Neck Cancer Receiving Cisplatin and Radiation Therapy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Financial Sponsor requested termination
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Cleveland BioLabs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 209611; NCI-2012-02140 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-11-13; First posted 2012-11-19 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Mucositis; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Stage III Squamous Cell Carcinoma of the Hypopharynx; Stage III Squamous Cell Carcinoma of the Larynx; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Squamous Cell Carcinoma of the Nasopharynx; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage III Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage III Verrucous Carcinoma of the Larynx; Stage III Verrucous Carcinoma of the Oral Cavity; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IVA Squamous Cell Carcinoma of the Larynx; Stage IVA Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVA Squamous Cell Carcinoma of the Oropharynx; Stage IVA Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVA Verrucous Carcinoma of the Larynx; Stage IVA Verrucous Carcinoma of the Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Larynx; Stage IVB Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Oropharynx; Stage IVB Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVB Verrucous Carcinoma of the Larynx; Stage IVB Verrucous Carcinoma of the Oral Cavity; Stage IVC Squamous Cell Carcinoma of the Larynx; Stage IVC Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVC Squamous Cell Carcinoma of the Oropharynx; Stage IVC Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVC Verrucous Carcinoma of the Larynx; Stage IVC Verrucous Carcinoma of the Oral Cavity; Tongue Cancer
MeSH Terms: conditions — Mucositis; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — CBLB502; Radiotherapy, Intensity-Modulated; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (entolimod, IMRT, cisplatin) (Experimental): Patients undergo IMRT 5 times per week for 7 weeks, receive cisplatin IV once weekly for 7 weeks, and entolimod SC on days 1, 8, 15, 22, 29, 36, and 43.
  Interventions: Drug: entolimod; Radiation: intensity-modulated radiation therapy; Drug: cisplatin; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: entolimod — Given SC
  Other Names: CBLB502; TLR5 agonist CBLB502; toll-like receptor 5 agonist CBLB502
Radiation: intensity-modulated radiation therapy — Undergo IMRT
  Other Names: IMRT
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of entolimod in treating patients with stage III-IV or recurrent head and neck cancer. Biological therapies, such as entolimod, may stimulate the immune system in different ways and stop tumor cells from growing. Entolimod may also prevent side effects caused by chemotherapy with cisplatin and radiation therapy. Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving entolimod together with cisplatin and radiation therapy may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the Phase II dose of CBLB502 (entolimod) when given as weekly injections during irradiation with cisplatin, for patients with poor prognosis advanced squamous cell carcinomas of the head and neck receiving chemoradiotherapy.

SECONDARY OBJECTIVES:

I. To describe the adverse event (AE) profile and the dose limiting toxicities of CBLB502 when administered weekly in combination with cisplatin and radiation therapy.

II. To determine the maximally tolerated dose (if observed) of CBLB502 in combination with cisplatin and radiation therapy.

III. To describe the pharmacokinetics (PK) of CBLB502 when administered in combination with cisplatin.

IV. To describe the pharmacodynamics (PD) of CBLC502 by examining plasma levels of various cytokines, including filgrastim (granulocyte-colony stimulating factor [G-CSF]), interleukin (IL)-6, IL-8, IL-10, and tumor necrosis factor-alpha (TNF-α).

V. To describe any clinical activity of CBLB502 in the form of mitigation of mucositis.

VI. To describe the response rate to chemoradiotherapy in combination with CBLB502.

OUTLINE: This is a dose-escalation study of entolimod.

Patients undergo intensity-modulated radiation therapy (IMRT) 5 times per week for 7 weeks, receive cisplatin intravenously (IV) once weekly for 7 weeks, and entolimod subcutaneously (SC) on days 1, 8, 15, 22, 29, 36, and 43.

After completion of study treatment, patients are followed up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of squamous cell carcinoma (stage III - IV) of the nasopharynx, oropharynx, oral cavity, paranasal sinuses, larynx, hypopharynx; the tumor must be human papillomavirus (HPV) negative or the patient should have a greater than 10 packs year smoking history; OR need for post-operative concurrent chemoradiotherapy (extracapsular extension, positive surgical margin, more than 1 lymph node positive, stage III - IV disease, perineural invasion, vascular tumor embolus) for histologically proven squamous cell carcinoma of the paranasal sinuses, nasopharynx, larynx, hypopharynx, with extension to structures of the oropharynx
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Induction chemotherapy (up to 3 cycles of cetuximab/taxanes/platinum based regimens) is allowed
* Patients or their legal representatives must be able to comprehend and provide written informed consent
* Absolute neutrophil count => 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit normal (ULN)
* Calculated creatinine clearance >= 60 mL/min (Cockcroft-Gault equation)
* 12-Lead Electrocardiogram (ECG) with normal tracing or non-clinically significant changes that do not require medical intervention
* Bazett's corrected QT (QTcB) interval < 470 msec at any timepoint prior to receiving the first dose of study drug (mean of replicate values, correction per institutional standard) and no history of Torsades des Pointes or other symptomatic QTcB abnormality
* Absence of orthostatic hypotension
* Patients must be sufficiently recovered from induction chemotherapy to allow initiation therapy

Exclusion Criteria:

* Women of childbearing potential who do not have a negative serum pregnancy test performed within 7 days prior to the start of study drug
* Male and female patients of child-bearing potential who do not agree to use double-barrier contraceptive measures, oral contraception, or avoidance of intercourse during the study and for 90 days after last investigational drug dose received
* Contraindication to full course chemoradiotherapy with cisplatin
* Previous treatment with a toll-like receptor 5 (TLR5) agonist
* Presence of neutralizing antibodies to CBLB502
* Patients with an active infection or with a fever >= 38.5ºC within 3 days of the first scheduled day of dosing; patients who are registered but develop a fever of >= 38.5ºC may remain in the study if the fever abates prior to the expiration of the screening procedures; if the screening procedures have expired, the patient may be re-screened once afebrile
* Patients with a history of significant cardiovascular, neurological, endocrine, gastrointestinal, respiratory or inflammatory illness that could preclude their participation in the study, pose an undue medical hazard or interfere with the interpretation of the study results, including, but not limited to, patients with congestive heart failure (New York Heart Association [NYHA] class 3 or class 4); unstable angina; cardiac arrhythmia; recent (within the preceding 6 months) myocardial infarction or stroke; hypertension requiring > 2 medications for adequate control; diabetes mellitus with > 2 episodes of ketoacidosis in the preceding 12 months; chronic obstructive pulmonary disease (COPD) requiring > 2 hospitalizations in the preceding 12 months
* Patients with a history of, or known autoimmune disease, but not limited to systemic lupus erythematosus, rheumatoid arthritis, systemic sclerosis, ankylosing spondylitis, sarcoidosis, vasculitis, Wegener's granulomatosis, Hashimoto's thyroiditis, ulcerative colitis, Crohn's disease, Goodpasture's disease, multiple sclerosis, etc.
* Patients with any other medical, psychiatric or social condition that would preclude their participation in the study, pose an undue medical hazard, interfere with the conduct of the study or interfere with interpretation of the study results
* Patients taking sucralfate, palifermin or amifostine
* Patients receiving hematopoietic growth factors
* Patients currently taking, or who have taken within 30 days of the initiation of protocol therapy, any immunomodulatory therapy, including pharmacologic doses of glucocorticoids (topical and inhalation glucocorticoids are permitted), azathioprine, methotrexate, interferon-alpha, interferon-beta, interluekin-2, etanercept, infliximab, tacrolimus, cyclosporine, mycophenolic acid, etc
* Patients with a history of hypersensitivity reactions to any of the components of CBLB502 or cisplatin
* Women who are pregnant or lactating or who are planning on becoming pregnant during the study or for 90 days after completion of the study
* Patients who have received an investigational therapy within 4 weeks of signing the informed consent for the current study
* Patients with a history of, patients who were treated for, or patients who are suspected of having, hepatitis B, and hepatitis C or human immunodeficiency virus (HIV); patients suspected of having any of these conditions should undergo appropriate evaluations prior to being enrolled in the study
* Surgery with significant defect or flap in the oral cavity
* Poor dentition or ill-fitting dental appliances (can be enrolled if this can be corrected by a dentist prior to start of radiation therapy)
* Presence of other medical conditions causing mucositis (e.g., rheumatologic, gastroesophageal reflux, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Adverse events defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related graded according to Common Toxicity Criteria for Adverse Events (CTCAE) version 4.0 | Up to 3 months after completion of study treatment
  Summarized descriptively by time point (mean, standard deviation). All safety analyses will be presented by dose cohort and overall as well as examined for relation to demographic parameters (i.e., gender, weight, body surface area [BSA]) and covariance or dependence on PK, PD, or presence of anti-entolimod antibodies at baseline and/or the development of entolimod antibodies.
PK of entolimod when administered in combination with cisplatin and radiation therapy | Predose, and at 2, 4, 6, 8, and 12 (+/- 2) hours postdose on Day 1
  A population PK model will be developed utilizing the PK time points collected and used to estimate individual areas under the curve (AUCs) or clearance (CL) of entolimod. The effect of patient factors, such as demographics and ECOG status, on entolimod PK will be evaluated by the model to help explain the interpatient variability in PK. Entolimod AUC, as well as the observed Crnax, will then be tested for association changes in cytokine levels, such as G-CSF, IL-6, IL-8, IL- 10 and TNF-alpha.
The percentage of patients with mucositis, measured using the World Health Organization (WHO) mucositis global severity score and the oral mucositis daily questionnaire (OMDQ) | Up to 3 months after completion of study treatment
  The percentage of patients with mucositis will be tabulated overall and by dose level.

CONTACTS AND LOCATIONS:
Overall Officials: Anurag Singh, Principal Investigator — Roswell Park Cancer Institute